CLINICAL TRIAL: NCT00413673
Title: Initial Evaluation of Photorefractive Keratectomy in U.S. Army Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU # 2335-99
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2007-11

CONDITIONS: Myopia
Keywords: Naturally occurring low to moderate myopia, with or without low levels of astigmatism in U.S. Army personnel
MeSH Terms: conditions — Myopia

ARMS (1):
- 1 (Experimental): PRK
  Interventions: Procedure: PRK

INTERVENTIONS:
Procedure: PRK — PRK

SUMMARY:
The objective of this study is to conduct a prospective clinical trial to evaluate the safety and efficacy fo the VISX Excimer Laser system for the treatment of naturally occurring low to moderate myopia, with or without low levels of astigmatism, in U.S. Army personnel.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Normal, healthy active adults with access to medical care at Walter Reed Health Care System.
* Age 21 years or older.
* Spherical equivalent of the manifest refractive error between -1.0 to -6.0 diopters (D), inclusive, with no more than 3.0D of cylinder. The absolute value of the cylinder (expressed in minus cylinder) will be limited such that the short axis of the elliptical ablation will be no smaller than 4.9mm. The following specifies the maximum cylinder for a given spherical component of the manifest refraction:

Spherical component / Maximum cylinder

* 1.0D / -0.5D
* 2.0D / -1.0D
* 3.0D / -1.5D
* 4.0D / -2.0D
* 5.0D / -2.5D
* 6.0D / -3.0D
* Corrected vision of at least 20/20
* Soft contact lens users must havE removed their lenses at least two weeks prior to baseline measurements.
* Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least four weeks prior to baseline measurements. At least two weekly manifest refractions and keratometry measurements will be required in this interval. The last two measurements must not vary by more than 0.50D in any meridian.
* Patients undergoing orthokeratology must have their lenses removed at least 6 months prior to the baseline examination. At least two monthly manifest refractions and keratometry measurements taken after the third month out of lenses must not vary by more than 0.50D in any meridian.
* Refractive stability must be documented by previous refractions. Spherical and cylindrical portion of the manifest refraction must not have varied by more than 0.50D over the previous 12 months.
* Exhibits strong motivation for keeping the follow-up visits.
* Available for evaluation at Walter Reed during the two-year follow-up period.
* Service members must have their command approval to participate in the study.
* Access to transportation to meet follow-up requirements.

Exclusion Criteria:

* Residual, recurrent or active ocular diseases or corneal abnormalities in either eye such as iritis, uveitis, keratoconjunctivitis sicca, herpetic keratitis, vernal conjunctivitis, lagophthalmos, corneal scarring, glaucoma, previous steroid responder, occludable chamber angles, visually significant cataracts.
* Either one or both eyes suffering from chronic dryness.
* Taking any systemic medications that may affect wound healing such as corticosteroids or antimetabolites.
* Patient corneal neovascularization within one mm of the ablation zone.
* History of any previous eye surgery, including previous refractive surgery.
* Best corrected visual acuity of less than 20/20.
* Progressive myopia or keratoconus.
* Any systemic disease that may affect wound healing, such as connective tissue disorders (rheumatoid arthritis, systemic lupus erythematosus, etc.), diabetes, or severe atopic disease.
* Any physical or mental impairment that would preclude participation in any of the examinations.
* For contact lens users there must be no evidence of contact lens corneal warpage on computerized topography.
* Currently on flight status or projected to be on flight status within ten years.
* Pregnant or breast-feeding an infant. Women of childbearing age must take a urine blood pregnancy test before starting this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2001-08; Study Completion 2008-03

PRIMARY OUTCOMES:
safety and efficacy of PRK | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: KRAIG S. BOWER, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Center For Refractive Surgery, Washington D.C., District of Columbia, United States